CLINICAL TRIAL: NCT04394442
Title: Use of Hydroxychloroquine in Patients With COVID-19: A Randomized Controlled Clinical Trial
Brief Title: Hydroxychloroquine in COVID-19 Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samah Lutfy (Other Government)
Responsible Party: Sponsor-Investigator, Samah Lutfy, Assistant professor of chest diseases, Zagazig University
Organization: Zagazig University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNH1352020
Record Dates: First submitted 2020-05-17; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxycholoroquine group (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Control group (No Intervention)

INTERVENTIONS:
Drug: Hydroxychloroquine — 400mg BD first day then 200 mg BD for 5 days
  Arms: Hydroxycholoroquine group

SUMMARY:
Many reports argued about the possible beneficial effects of Hydroxychloroquine in treating COVID-19 patients and this study was designed to investigate this claim

ELIGIBILITY:
Inclusion Criteria:

Confirmed cases of SARS-CoV-2 by PCR

Exclusion Criteria:

less than 18 years old known hypersensitivity to the drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-21 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
time to viral clearance | 21 days after patients randomization
  PCR will be done every 72 h day till 2 consecutive negative PCR tests(24h apart) which is the viral clearance.The time between randomization and viral clearance is the viral clearance time
% of mortality | 60 days after randomization
  total number of deaths divided by total number of the group

SECONDARY OUTCOMES:
Length of stay | 60 days after randomization
  time from patients randomization till discharge
time to be afebrile | 60 days after randomization
  time from randomization till day of fever subsiding
need for mechanical ventilation | 60 days after randomization
  %of deteriorated patients necessitates mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- SNH, Mecca, Saudi Arabia